CLINICAL TRIAL: NCT06725459
Title: Assessing the Application of Closed Incision Negative Pressure Wound Therapy to Reduction Mammaplasty
Brief Title: NPWT Reduction Mammaplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00007266
Record Dates: First submitted 2024-11-15; First posted 2024-12-10 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Healthy; Macromastia; Negative Pressure Therapy; Mammaplasty; Wound Healing
Keywords: mammaplasty; macromastia; breast reduction; negative pressure therapy
MeSH Terms: conditions — Gigantomastia

STUDY DESIGN:
Intervention Model Description: The Prevena Restor Bella Form™ wound vacuum will be applied to the reduction mammaplasty incision as directed for up to 7 days postoperatively. Prevena Restor Bella Form™ is a ciNPWT management system. ciNPWT management systems apply negative pressure to the incision and structurally stabilize the surrounding tissues.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Prophylactic ciNPWT (Experimental): Participants in this arm will receive the prophylactic closed incision negative pressure wound therapy (ciNPWT) on one breast following reduction mammaplasty. The ciNPWT will be applied for up to 7 days postoperatively to promote wound healing and prevent complications.
  Interventions: Device: Prophylactic ciNPWT
- Standard Adhesive Dressing (Active Comparator): Participants in this arm will receive the standard adhesive strip dressing (Prineo Ethicon NJ) on the other breast following reduction mammaplasty. The standard dressing will be used as a control to compare postoperative outcomes against the ciNPWT.
  Interventions: Other: Standard Adhesive Dressing

INTERVENTIONS:
Device: Prophylactic ciNPWT — The prophylactic closed incision negative pressure wound therapy (ciNPWT) will be applied to one breast for up to 7 days postoperatively to promote wound healing and prevent complications.
  Arms: Prophylactic ciNPWT
Other: Standard Adhesive Dressing — The standard adhesive strip dressing will be applied to one breast immediately after surgery. It provides a protective covering for the wound during the initial healing phase and is the standard of care for incision management.
  Arms: Standard Adhesive Dressing

SUMMARY:
In this prospective, randomized, split-body control trial, we aim to compare complications, patient-reported outcomes, and cost differentials following reduction mammaplasty with prophylactic closed incision negative pressure wound therapy versus standard adhesive dressing.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Age 18 years or older
* Scheduled to undergo bilateral reduction mammaplasty with a Wise pattern (anchor) incision and a superomedial, inferior, or central mound pedicle at MedStar Georgetown University Hospital or MedStar Good Samaritan Hospital
* Able to comply with study procedures and follow-up visits

Exclusion Criteria:

* Younger than 18 years of age
* Biologically male patients
* Scheduled to undergo unilateral breast mammaplasty
* Currently pregnant or lactating
* Use of steroids or other immune modulators known to affect wound healing
* Current smokers who have not paused for a minimum of 4 weeks prior to surgery
* History of breast cancer
* History of oncologic or reconstructive breast surgery
* History of radiation to the breast
* History of chemotherapy or hormone therapy
* Tattoos in the area of skin incision
* Skin conditions known to affect wound healing or scarring of the breast (e.g., cutis laxa)
* Significant history of scar problems (e.g., hypertrophic scarring or keloids) post-surgical incisions with active bleeding
* Exposure of blood vessels, organs, bone, or tendon at the base of the reference wound
* Known allergies to product components (e.g., medical or NPWT tape)
* Unable to comply with NPWT requirements, including those unable to present for postoperative follow-up
* Lactating at the time of surgery
* Require deviation from standard operative or closure techniques (e.g., staples, free nipple grafts)
* Considered part of a vulnerable population (adults unable to consent, infants, children, teenagers, pregnant women, prisoners)
* Experience intraoperative complications due to surgical complications not related to the NPWT instrumentation (e.g., expanding hematoma)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Wound Complications | 30 days postoperatively
  The primary outcome measure is the incidence of postoperative wound complications within 30 days following reduction mammaplasty. This includes surgical wound dehiscence, delayed wound healing, and surgical site infections (SSIs).

SECONDARY OUTCOMES:
Patient-Reported Pain (VAS) | Immediate postoperative period, 1 week postoperatively, and 3 months postoperatively
  Patient-reported pain will be assessed using the Visual Analog Scale (VAS) with scores ranging from 0 (no pain) to 10 (maximal imaginable pain).
Scar Quality (POSAS) | 1 month and 3 months postoperatively
  Scar quality will be assessed using the Patient and Observer Scar Assessment Scale (POSAS) at 1 and 3 months postoperatively. The scale ranges from 6 (normal skin) to 60 (worst imaginable scar).
Patient Satisfaction with Breasts (BREAST-Q) | Preoperative baseline, 1 week postoperatively, 1 month postoperatively, 3 months postoperatively, and 6 months postoperatively
  Patient satisfaction with their breasts will be measured using the standardized BREAST-Q 2.0© questionnaire at the preoperative consultation, and at 1 week, 1 month, 3 months, and 6 months postoperatively.
Cost Differential: Dressing-Related Costs | Through study completion, an average of 6 months
  Costs associated with dressings will include the unit price of ciNPWT and standard adhesive dressings and healthcare professional time for application and removal.
Cost Differential: Healthcare Resource Use | Through study completion, an average of 6 months
  Healthcare resource use will include hospital stay durations, additional procedures for managing complications, and any unplanned follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth L Fan, MD, Principal Investigator — MedStar Georgetown University Hospital
Locations (1):
- Medstar Georgetown University Hospital, Washington D.C., District of Columbia, United States